CLINICAL TRIAL: NCT06286969
Title: Clinical Study on the Treatment of Lumbar Muscle Strain by Intensive Multi-acupuncture Method Based on the Principle of "Tendons Disease Pain-point Needling".
Brief Title: Clinical Study on Intensive Multi-acupuncture in the Treatment of Lumbar Muscle Strain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Xinnan (Other)
Responsible Party: Sponsor-Investigator, Xu Xinnan, medical student, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZSLL-ZN-2024-007-01
Record Dates: First submitted 2024-02-24; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Lumbar Muscle Strain
MeSH Terms: conditions — Sprains and Strains | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intensive multi-acupuncture method group (Experimental): The needle entry points of the lower row are straight punctures that penetrate the muscle attachments along the medial superior margin of the posterior superior iliac spine, the medial margin of the sacroiliac joint, and a portion of the lateral iliac crest of the lumbar triangle. The entry point of the upper row of needles was made oblique, and then small lifting insertion, respectively, reached and penetrated the anterior border muscle attachments. Then subperiosteal stabbing along the bone surface was used to penetrate 1.5cm forward and downward, and the needle was retained for 15min. The needle was left in place for 15 min, and for the second puncture, the entry point was chosen to be in the middle of the two longitudinal entry points of the first puncture. The rest of the operation was unchanged. Repeat the above operation for the last 3 treatments. The treatment is performed twice a week for a total of 5 treatments.
  Interventions: Procedure: acupuncture
- normal needling group (Experimental): The points were selected with reference to the 2006 National Standard of the People's Republic of China (GB/T 12346-2006), "Acupoint Names and Localization". The patients were placed in the prone position, the acupoints were sterilized with 75% alcohol, and the needles were inserted vertically with the conventional needling method, to the extent that there was a sensation of acidity, numbness, heaviness, distension, or radiating to the surroundings, and the needles were left in place for 15 min. The treatments were carried out twice a week for a total of five treatments.
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — The needles are inserted into the subject in a certain way to stimulate specific parts of the body to treat the disease.

SUMMARY:
Acupuncture is widely used as a routine treatment for lumbar muscle strain. The aim of this randomized controlled trial is to evaluate the effectiveness of the intensive multi-acupuncture method. This trial will include 108 patients with lumbar muscle strain injury from two outpatient clinics. All participants will be randomized in a 1:1 ratio to the intensive multi-acupuncture method group and the normal needling group. Outcomes will be assessed before the intervention, after one treatment, after five treatments, and at follow-up 2 weeks after the end of treatment. The primary outcome indicator will be the clinical efficacy evaluation criteria, and the secondary outcome indicators will be the pain visual analog scale (VAS) score, the Japanese Orthopaedic Association Assessment Treatment Score (JOA) score, the lumbar joint mobility measurement scale, and the Modified Ashworth Grading Scale. This study will provide evidence as to whether the intensive multi-acupuncture method is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

1.Meet the above Chinese and Western medicine diagnostic criteria; 2.18 years old ≤ age ≤ 70 years old, gender is not limited; 3.The duration of the disease is more than 3 months, no other treatment has been received in the last month, and the VAS score is ≥4 at the time of participating in the treatment; 4.Voluntarily cooperate with the examination and treatment, and sign the Informed Consent Form.

Exclusion Criteria:

1. Those with severe cardiac, hepatic and renal insufficiency and those with bleeding tendency;
2. Previous history of lumbar spine surgery, spinal cauda equina tumor, lumbar spondylolisthesis, lumbar spinal stenosis, scoliosis deformity, tumors and other diseases caused by low back pain;
3. Women who are in the period of pregnancy or breastfeeding should not perform acupuncture treatment;
4. Those who have needle-sickness, blood-sickness and so on;
5. Those who have cognitive impairment and cannot complete the relevant scale assessment independently or under the guidance of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
clinical efficacy evaluation criteria | Outcomes will be assessed after one treatment, after five treatments, and at follow-up 2 weeks after the end of treatment.
  It was evaluated according to the efficacy standard of lumbar muscle strain injury in the Guidelines for Clinical Research of New Chinese Medicines, and the JOA index was used as the benchmark:
  Efficacy index (N) = [(pre-treatment score - post-treatment score) ÷ pre-treatment score] × 100%
  * cure: the patient does not feel obvious back pain and other discomforts, N ≥ 90%
    * Effective: Effective: low back pain is significantly relieved, 60% ≤ N < 90% ③ Effective: lower back pain is relieved, 30%≤N<60%. ④ Ineffective: the patient's low back pain is not relieved, N<30%. Total effective rate (%) = [(number of cured + number of effective + number of effective) ÷ number of cases in each group] × 100%.

SECONDARY OUTCOMES:
Pain visual analog scale (VAS) score | Outcomes will be assessed before the intervention, after one treatment, after five treatments, and at follow-up 2 weeks after the end of treatment.
  The visual analogue scale (VAS) is used for pain assessment. The basic method is to use a traveling scale of about 10 cm in length, with 10 scales on one side and "0" and "10" scores at each end, with 0 indicating no pain and 10 representing the most severe pain that is intolerable.
Japanese Orthopaedic Association Scores | Outcomes will be assessed before the intervention, after one treatment, after five treatments, and at follow-up 2 weeks after the end of treatment.
  JOA refers to the Japanese Orthopaedic Association Assessment Treatment Score, which is primarily used to evaluate functional impairment in the human body.The total JOA score ranges from a maximum of 29 to a minimum of 0. The lower the score, the more pronounced the functional impairment. Lower scores indicate more significant dysfunction.
Lumbar Joint Mobility Measurement Scale | Outcomes will be assessed before the intervention, after one treatment, after five treatments, and at follow-up 2 weeks after the end of treatment.
  The lumbar mobility test is an examination of the mobility of the lumbar region. The tester is asked to perform forward flexion, backward extension, lateral flexion, and rotational movements to assess the degree of limitation of lumbar mobility.
Improvement of the Ashworth Rating Scale | Outcomes will be assessed before the intervention, after one treatment, after five treatments, and at follow-up 2 weeks after the end of treatment.
  The Modified Ashworth Grading Scale assesses the degree of spasticity of the lumbar muscles by measuring muscle tone during exercise.